CLINICAL TRIAL: NCT06075303
Title: Dynamic Assessment of Phonological Disorders: Part 1 Assessment & Part 2 Treatment
Brief Title: Dynamic Assessment of Phonological Disorders
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Montana (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: 186-11
Record Dates: First submitted 2023-10-03; First posted 2023-10-10 (Actual); Last update posted 2023-10-10 (Actual); Status verified 2023-10

CONDITIONS: Speech Sound Disorder
Keywords: phonology, delay, disorder, speech
MeSH Terms: conditions — Speech Sound Disorder; Speech

STUDY DESIGN:
Intervention Model Description: Children will engage in 4 weeks of treatment on easier targets and 4 weeks of treatment on harder targets. The order (easier first or harder first) will be counterbalanced across participants.
Who Masked: Participant
Masking Description: The participating children will not be aware of the targets identified as "easier" or "harder"
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Easier Targets (Experimental): All participants will participate in a modified Cycles approach where speech targets are worked on for a short period of time and switched within a cycle. During the Easier Targets arm, children will work on target sounds that are "easier" based on their pre-treatment scores of 8, 9, 10, or 11 on the Glaspey Dynamic Assessment of Phonology. Children will complete 8 sessions in this arm that are each 50-minutes long and occur two times per week with each target addressed for 2 sessions.
  Interventions: Behavioral: Modified Cycles
- Harder Targets (Experimental): All participants will participate in a modified Cycles approach where speech targets are worked on for a short period of time and switched within a cycle. During the Harder Targets arm, children will work on target sounds that are "harder" based on their pre-treatment scores of 15, 14, 13, or 12 on the Glaspey Dynamic Assessment of Phonology. Children will complete 8 sessions in this arm that are each 50-minutes long and occur two times per week with each target addressed for 2 sessions.
  Interventions: Behavioral: Modified Cycles

INTERVENTIONS:
Behavioral: Modified Cycles

SUMMARY:
The goal of this clinical trial is to learn about (1) how speech skills can be measured and how various tests give speech therapists different types of information for children with speech sound disorder, and (2) whether changes occur in the amount of help children need when they work on easier sounds or harder sounds during treatment. The main questions this study aims to answer are: (1) what does one type of test (dynamic assessment) tell us about speech skills compared to another type of test (static assessment), and (2) does practice of easier or harder sounds show differences in progress. Participants will complete 16 sessions of speech treatment called "modified cycles treatment", and will complete several speech and language tests before, during, and after treatment by pointing to pictures, and saying sounds, words, and sentences.

DETAILED DESCRIPTION:
The Glaspey Dynamic Assessment of Phonology (GDAP) (Glaspey, 2006; Glaspey & Stoel-Gammon, 2007) was initially developed because children with speech-sound delays make very slow progress in speech therapy and it is difficult to document change in short periods of time using traditional methods of assessment. The traditional methods rely on picture-naming tasks and the child is not given any assistance in speech productions. The lack of assistance often results in a floor effect in the documentation of change and progress. Without good documentation of change, speech-language pathologists are left uncertain about the efficacy of the treatment that they are administering. The GDAP is unique because it assesses change based on dynamic assessment; children are systematically given assistance in the production of speech sounds. When administering the GDAP, clinicians rate each sound on a 15-point ordinal scale that represents the number of cues and assistance that could be used to assist the child in sound production. Progress is documented as children need less support over time and their scores decrease. This study compares the GDAP with a traditional single-word measure. This study also has an extension to use the GDAP to select easier or harder targets during treatment, and monitor children's progress across measures over 8 weeks of modified cycles treatment. The treatment will include 16 sessions of therapy with two 50-minute sessions per week. The treatment approach that will be used is called "Cycles" and involves practicing a different speech sound each week (Rudolf & Wendt, 2014). The sounds that are practiced will be individualized to each child's needs, with harder sounds taught during four of the weeks and easier sounds taught during four of the weeks. The order will be counter-balanced across participants.

ELIGIBILITY:
Inclusion Criteria:

* monolingual English speakers;
* scores in the mild to profound range for phonological disorder based on the Hodson Assessment of Phonological Patterns (Hodson, 2004);
* scores above 9th percentile on receptive language and cognitive abilities based on measures from the Preschool Language Scale-4 (PLS-4) (Zimmerman, Steiner, & Pond, 2002) and the Peabody Picture Vocabulary Test (PPVT) (Dunn & Dunn, 1997);
* perform adequately on a structural-functional examination adapted from the Oral and Speech Motor Control Protocol (Robbins & Klee, 1987) and Motor Speech Examination (Strand & McCauley, 1999);
* exhibit voice and fluency skills within normal limits,
* pass a hearing screening adequate for understanding speech.

Exclusion Criteria:

* will not exhibit the prime characteristics of developmental apraxia of speech and/or dysarthria

Ages: 3 Years to 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 4 (Actual)
Dates: Start 2011-10-04 (Actual); Primary Completion 2012-05-11 (Actual); Study Completion 2012-05-11 (Actual)

PRIMARY OUTCOMES:
Glaspey Dynamic Assessment of Phonology (GDAP) | Prior to treatment, after four weeks of treatment, and again after eight weeks.
  The GDAP is an evaluation of speech sounds when given help while talking about pictures.
  The child is asked to say all sounds by themselves, in words, or in sentences. The child is given verbal modeling and instructions to help him/her say the sounds correctly to the highest level possible (i.e. sentences without any model).

SECONDARY OUTCOMES:
Static Assessment of Single Words | Prior to treatment, after four weeks of treatment, and again after eight weeks.
  Evaluation of speech sounds in words using pictures. The child will be shown 50-80 picture cards and asked to say the pictures. There pictures feature sounds that may be in error by the child.

CONTACTS AND LOCATIONS:
Overall Officials: Amy M Glaspey, Ph.D., Principal Investigator — University of Montana

IPD SHARING:
Plan to Share IPD: No